CLINICAL TRIAL: NCT06496074
Title: Sex-Specific Heart Rate Variations in Predicting Outcomes of Head-Up Tilt Tests in Syncope Patients
Brief Title: Heart Rate Variation in Females Predicts Tilt Test Results
Status: Active, not recruiting | Type: Observational
Sponsor: Federal University of Piaui (Other)
Responsible Party: Principal Investigator, Carlos Eduardo Batista de Lima, MD, PhD, Professor of Medicine (Cardiology), Federal University of Piaui
Other Study IDs: FUPiaui_tilt_test
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Syncope, Vasovagal
Keywords: Vasovagal syncope; Tilt-table test; Heart rate variation; Blood pressure; Hemodynamics
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive head-up tilt test: Patients who underwent to head-up tilt test (HUTT) and met criteria for positive exam according to the defined in guidelines.
  Interventions: Diagnostic Test: Head-up Tilt Test
- Negative head-up tilt test: Patients who underwent to head-up tilt test (HUTT) and did not met criteria for positive exam according to the defined in guidelines.
  Interventions: Diagnostic Test: Head-up Tilt Test

INTERVENTIONS:
Diagnostic Test: Head-up Tilt Test — Two protocols for the head-up tilt test (HUTT) are used in our center and in the collaborating centers: (1) passive or prolonged inclination protocol [40 minutes], (2) mixed protocol: passive phase [first 20 minutes] plus nitrate-provoked phase [last 20 minutes], with the use of 1.25 mg sublingual isosorbide dinitrate. All patients are submitted to 10 minutes of rest in the supine position at zero degree before the tilt phase of the HUTT. During this period, HR and systolic (SBP) and diastolic (DBP) measurements are obtained every 2 minutes. After this phase, the table is tilted at an angle of 70° with measurement of SBP / DBP and HR every minute. Patients older than 60 years are routinely investigated for carotid sinus hypersensitivity by carotid sinus massage during the passive phase of the HUTT. The exam is considered positive according to the criteria defined in guidelines.

SUMMARY:
Head-up tilt test (HUTT) is widely used to evaluate patients with unexplained syncope, but data on clinical predictors of HUTT results are limited. The investigators aim to evaluate heart rate (HR) variations and blood pressure (BP) changes associated with the HUTT results and the difference according to the gender. For this, a cross-sectional study will be performed with patients attended with unexplained syncope submitted to HUTT (70-degree angle), from January/2011 to April/2015. The investigators will analyze BP changes and Receiver-Operating Characteristics (ROC) curves for the maximum interval in HR variation from the first minute to tenth minute (delta-HR 10) after tilting. The significance level will be considered at 5%.

DETAILED DESCRIPTION:
The protocols for the HUTT are passive or prolonged inclination protocol [40 minutes] and mixed protocol: passive phase [first 20 minutes] plus nitrate-provoked phase [last 20 minutes], with the use of 1.25 mg sublingual isosorbide dinitrate. Blood pressure (BP) measurements will be obtained manually with the Welch Allyn® DS44-11BR, Durashock sphygmomanometer and heart rate (HR) data will be obtained continuously by cardiac monitoring in a conventional 12-lead ECG-PC TEB® surface electrocardiogram with automatic measurements certified by Brazilian National Standards/International Electrotechnical Commission (NBR/IEC) 60601-2-51 and registration number with Brazilian Health Regulatory Agency (ANVISA): 10265690026. All patients will be submitted to 10 minutes of rest in the supine position at zero degree before the tilt phase of the HUTT. During this period, HR and systolic (SBP) and diastolic (DBP) measurements will be obtained every 2 minutes. After this phase, the table is tilted at an angle of 70° with measurement of SBP / DBP and HR every minute. Patients older than 60 years are routinely investigated for carotid sinus hypersensitivity by carotid sinus massage during the passive phase of the HUTT. The exam is considered positive according to the criteria defined in guidelines. The variables analyzed are: age; sex; symptoms prior to examination including syncope, near-syncope and others including dizziness, palpitations and suspected dysautonomia; The maximum heart rate (HR) interval variations present from the rest phase up to the first minute (HR Delta 1min) and from the first minute up to the tenth minute (HR Delta 10min) in tilt phase are documented. The interval changes in systolic and diastolic blood pressure measurements are obtained from the last measurement of the rest phase up to the first minute in tilt phase. For statistical analysis, the Chi-square test will be used to verify the dependence or independence of variables considered by evaluating the association between qualitative variables. The t-Student test will be used to evaluate the differences between the means of the two groups. The Mann-Whitney test (Wilcoxon rank-sum test) will be used to compare two unpaired groups verifying whether or not they belong to the same population and whose requirements for applying the t-student test are not met. For the definition of the cutoff points of variations in HR, the ROC curves will be constructed for the HR delta 1 min and HR delta 10 min variables, evaluating the performance of these parameters and analyzing the sensitivity and specificity for their correlation with the positivity in the HUTT. Through the logistic regression model, the probability curves will be constructed for the HUTT positivity for the parameters of HR delta 1 min and HR delta 10 min and for the non-positivity in the HUTT in relation to the BP variation up to the second minute of the examination. The significance level will be considered at 5%. Statistical analysis will be performed using the Statistical Package for the Social Sciences (SPSS, version 18.0 for Windows).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients attended with a history of syncope submitted to head-up tilt test

Exclusion Criteria:

* Patients < 18 years old
* Patients without a history of true syncope
* Patients who did not submit to head-up tilt test
* Withdrawal of the consent form at the request of the patient or guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years old, male or female, with the presence of the inclusion criteria and without exclusion criteria, attended with a history of syncope submitted to head-up tilt test, between January 2011 and April 2015, by the Federal University of Piaui, Brazil in co-participation with the private sector including the Clinicardio and the ITACOR Hospital, specialized centers for diagnosis and treatment of the heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Positive diagnostic correlation | 30 days
  Positive diagnostic correlation of the data obtained in group 1 (positive head-up tilt test) in relation to group 2 (negative head-up tilt test).

SECONDARY OUTCOMES:
Blood pressure variation in the head-up tilt test | 30 days
  Accuracy, sensitivity, and specificity of blood pressure values as predictors of outcome in the head-up tilt test
Heart rate variation in the head-up tilt test | 30 days
  Accuracy, sensitivity, and specificity of heart rate values as predictors of outcome in the head-up tilt test

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Eduardo Batista Lima, MD, PhD, Principal Investigator — Federal University of Piaui
Locations (1):
- Carlos Eduardo Batista de Lima, Teresina, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No
I have no plan to share individual patient data with other researchers.

REFERENCES:
- [Derived] de Lima CEB, da Silva PAD, de Sa Nascimento SRA, de Freitas MVA, de Area Leao Moreira FG, Silvino VO, Ramos RM, Pereira Dos Santos MA. Sex-Specific heart rate acceleration as predictors of positive head-up tilt test outcomes in syncope patients. BMC Cardiovasc Disord. 2025 Nov 11;25(1):800. doi: 10.1186/s12872-025-05290-7. PMID 41219842